CLINICAL TRIAL: NCT03269773
Title: A Multi-center, Randomized, Double-blind, Parallel, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of FURESTEM-AD Inj. for Moderate to Severe Chronic Atopic Dermatitis
Brief Title: Safety and Efficacy of FURESTEM-AD Inj. in Patients With Moderate to Severe Chronic Atopic Dermatitis(AD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K0102
Record Dates: First submitted 2016-10-05; First posted 2017-09-01 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Stem cell; Cell therapy; skin disease; Umbilical cord Blood; UCB-MSC; hUCB-MSC; AD; furestem; dermatitis; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases; Dermatitis; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FURESTEM-AD Inj. (Experimental): hUCB-MSC 5.0x10^7 cells
  Interventions: Biological: FURESTEM-AD Inj.
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: FURESTEM-AD Inj. — 0.3mL of the following study drug is injected respectively into both upper arms, both thighs, and abdomen (total of 5 regions) as a single dose (total 1.5 mL).
  Treatment group: FURESTEM-AD® inj. 5.0 X 107 cells/1.5 mL
  Arms: FURESTEM-AD Inj.
Other: Placebo — 0.3mL of the following study drug is injected respectively into both upper arms, both thighs, and abdomen (total of 5 regions) as a single dose (total 1.5mL)
  Arms: Placebo

SUMMARY:
This is multi-center, randomized, double-blind, parallel, placebo-controlled phase III clinical trial to evaluate the efficacy and safety of FURESTEM-AD Inj. for moderate to severe chronic atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Of either gender, aged >=19
2. Atopic Dermatitis subjects who are coincident with Hanifin and Rajka diagnosis criteria
3. Chronic Atopic Dermatitis that has been present for at least 3 years
4. EASI>=12 at screening and baseline visit
5. IGA>=3, SCORAD index>=25, BSA >=10% of AD involvement at screegning and baseline visit
6. Subjects with documented record of inadequate response to the stable use of topical atopic dermatitis treatment within 24 weeks before participating in the study, or whom are inadvisable due to safety risks
7. Subjects who understand and voluntarily sign an informed consent form

Exclusion Criteria:

1. Subjects with medical history or surgery/procedure history
2. Subjects with diseases at the time of participation in this study (systemic infection, other serious skin disorders, pigmentation or extensive scarring in atopic dermatitis symptom region)
3. Subjects who need prohibited medication during clinical period
4. Pregnant, breast-feeding women or women who plan to become pregnant during this study
5. Subjects who currently participate in other clinical trial or participated in other clinical trial within 4 weeks
6. Any other condition which the investigator judges would make patient unsuitable for study participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
over 50% reduction ratio of Eczema Area and Severity Index (EASI) as contrasted with baseline value (EASI-50) | 12 week

SECONDARY OUTCOMES:
over 75% reduction ratio of Eczema Area and Severity Index (EASI) as contrasted with baseline value (EASI-75) | 12 week
Change and rafe of change in EASI index | 24weeks
Proportion of patients who Investigator's Global Assessment (IGA) score 0 or 1 | 24weeks
Proportion of patients who Investigator's Global Assessment (IGA) score 0 or 1, or reduced more than 2 points | 24weeks
over 50% reduction ratio of SCORing Atopic Dermatitis (SCORAD) INDEX as contrasted with baseline value (SCORAD-50) | 24weeks
Change and rafe of change in SCORAD index | 24weeks
Change and rafe of change in Body Surface Area (BSA) | 24weeks
Change in total serum Immunoglobulin E (IgE) | 24weeks
Change in Cytokine (TNF-a, Interleukin (IL)-4, IL-5, IL-6, IL-8, IL-13, IL-31, TARC (CCL17) and CCL 27 analysis) | 24weeks
Total number of use and consumed amount of rescue medicine | 24weeks

CONTACTS AND LOCATIONS:
Locations (11):
- South Korea (11):
  - Pusan National University Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Dongguk University Medical Center, Ilsan
  - Gachon University Gil Medical Center, Incheon
  - Catholic Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University Healthcare System, Seoul
  - Hanyang University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Undecided